CLINICAL TRIAL: NCT02234076
Title: A Study on the Efficacy of Virtual Reality Exposure Therapy (VRET) for Survivors of Childhood Sexual Abuse and War Related Trauma
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Erasmus Medical Center (Other)
Collaborators: Netherlands Organisation for Scientific Research (Other Government); Erasmus University Rotterdam (Other); Delft University of Technology (Other); University of Amsterdam (Other); PsyQ (Other); Reinier van Arkel Groep, Psychotraumacentrum Zuid-Nederland (Unknown)
Responsible Party: Principal Investigator, Ingmar Franken, Professor of Clinical Psychology, Erasmus Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CI1-12-S028-1
Record Dates: First submitted 2014-07-15; First posted 2014-09-09 (Estimated); Last update posted 2016-08-17 (Estimated); Status verified 2016-08

CONDITIONS: Posttraumatic Stress Disorder (PTSD); Depression
Keywords: Posttraumatic Stress Disorder; Depression; Treatment; VRET
MeSH Terms: conditions — Stress Disorders, Post-Traumatic; Depression | interventions — Virtual Reality Exposure Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- VRET (Experimental): Virtual Reality Exposure Therapy (VRET)
  The experimental treatment VRET is offered with the Multi-Modal Memory Restructuring System (3MR system) and a therapy manual. Participants can use this system at home. Note: The 3MR system is offered via a computer screen, no head-mounted display (HMD) equipment is used in this study.
  Interventions: Behavioral: VRET
- TAU (Active Comparator): Treatment As Usual
  Interventions: Behavioral: TAU

INTERVENTIONS:
Behavioral: VRET
  Other Names: Virtual Reality Exposure Therapy (VRET)
  Arms: VRET
Behavioral: TAU — Treatment as usual offered by the participating mental health care organisations
  Arms: TAU

SUMMARY:
Background: Childhood Sexual Abuse (CSA) and combat related war-trauma are associated with posttraumatic stress disorder (PTSD) and depression. PTSD is one of the most prevalent Diagnostic and Statistical Manual of Mental Disorders (DSM) axis 1 disorders for which psychotherapy is widely practiced. Depression is one of the most common co morbid disorders when PTSD is diagnosed. Exposure to the traumatic memories or cues of the traumatic event often plays an important role in reducing symptoms of PTSD. Also symptoms of PTSD and depression have been related to a reduced specificity in autobiographical memory.

Objective: This study will examine the efficacy of a Virtual Reality Exposure Therapy (VRET) in a CSA and war related trauma sample by comparing it with treatment as usual (TAU). It will also attempt to develop protocols to implement this new technology into clinical practice and collect data to develop a treatment progress prediction model.

Study design: A randomized controlled intervention study.

Study population: 144 individuals with memories of CSA or war related trauma and symptoms of PTSD and/or depression.

Intervention: VRET or TAU.

ELIGIBILITY:
Inclusion Criteria:

* principal diagnosis meeting DSM-IV criteria for PTSD and/or major depression following CSA or war related trauma
* between the ages of 18 and 70-years-old
* having sufficient fluency in Dutch to complete treatment and research protocol

Exclusion Criteria:

* current bipolar disorder
* current psychotic disorders
* current suicidality
* high dissociation level (Dissociative Experiences Scale (DES) cut-off score ≥ 40)

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 144 (Estimated)
Dates: Start 2014-10; Primary Completion 2016-10 (Estimated); Study Completion 2016-10 (Estimated)

PRIMARY OUTCOMES:
Posttraumatic Stress Disorder (PTSD) Checklist Diagnostic & Statistical Manual of Mental Disorders (DSM) 5 (PCL-5) to measure change from baseline self-reported symptoms of PTSD at the endpoint of the therapy (after completing 12 sessions) and follow-ups | At pre (baseline), post (after 12 therapy sessions with a minimum of 6 weeks and a maximum of 12 weeks), and follow-up (3 and 12 months post treatment) measurements
  The PCL-5 is a brief assessment that identifies the presence and symptom severity of PTSD. We use the PCL-5 to measure self-reported symptoms of PTSD.
Beck Depression Inventory-II (BDI-II) to measure change from baseline self-reported symptoms of depression at the endpoint of the therapy (after completing 12 sessions) and follow-ups | At pre (baseline), post (with a minimum of 6 weeks and a maximum of 12 weeks), and follow-up (3 and 12 months post treatment) measurements
  The BDI-II is a self-report questionnaire which measures the severity of depression in 21 statements, with four levels of increasing severity each. We use the BDI-II to measure self-reported symptoms of depression.

SECONDARY OUTCOMES:
The Outcome Questionnaire-45-2 (OQ-45-2) to measure change from baseline self-reported symptoms and well-being at the endpoint of the therapy (after completing 12 sessions) and follow-ups | At pre (baseline), post (with a minimum of 6 weeks and a maximum of 12 weeks) and follow up (3 and 12 months post treatment) measurements
  The OQ-45-2 is a questionnaire which measures well-being in three domains; symptom distress, interpersonal functioning and social role. We use the OQ-45-2 to measure improvement in well-being in participants as addition to the symptom checklists, and to make a useful translation of the research data into clinical practice.

OTHER OUTCOMES:
The Positive and Negative Affect Scale (PANAS) to measure change in self-reported emotional progress between therapy sessions | Two times per week during 6 weeks
  The PANAS is a self-report questionnaire to measure positive and negative affect. The PANAS measures specific feelings as 'interested', 'inspired' etc. We use the PANAS to measure change in these affects between therapy sessions.
The 9-item depression module of the Patient Health Questionnaire (PHQ) to measure self-reported emotional progress between therapy sessions | Two times per week during 6 weeks
  The PHQ is a self-report questionnaire which scores the nine DSM-criteria for depression. We use the PHQ to measure change in the nine primary depression symptoms between therapy sessions.
The shortened version (6 items) of the PCL-5 to measure change in self-reported emotional progress between therapy sessions | Two times per week during 6 weeks
  For general information PCL-5 see primary outcome section. We use 6 items of the PCL-5 to measure self-reported symptoms of PTSD between therapy sessions.
The self-report questionnaire Patient's acceptance of a Self-Management health system to asses participants' acceptance of the used technology | Post treatment (after 6 weeks)
  The self-report questionnaire Patient's acceptance of a Self-Management health system is a questionnaire to evaluate participants' acceptance of the technology used during the current study. Outcomes are important because they might implicate alterations to strengthen usability of the technology.
The Mini International Neuropsychiatric Interview 5.0.0. (MINI 5.0.0.) Dutch version to screen for Diagnostic and Statistical Manual of Mental Disorder (DSM)-IV diagnoses | At pre (baseline), post (after 12 therapy sessions with a minimum of 6 weeks and a maximum of 12 weeks), and follow-up (3 and 12 months post treatment) measurements
  The MINI 5.0.0. Dutch version is a semi-structured clinical interview to screen for DSM-IV diagnoses such as PTSD, major depression, bipolar disorder. We use the MINI 5.0.0. Dutch to check in- and exclusion criteria, and to determine change in diagnosis after therapy.

CONTACTS AND LOCATIONS:
Locations (3):
- Netherlands (3):
  - Reinier van Arkel Groep PTC ZN, 's-Hertogenbosch, North Brabant
  - Erasmus University Rotterdam, Rotterdam, South Holland
  - PsyQ, Rotterdam/The Hague, South Holland

REFERENCES:
- See also: Project website — http://ii.tudelft.nl/vesp/